CLINICAL TRIAL: NCT05411757
Title: A Single-Arm, Open-Label Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of IBR900 Cell Injection Combined With Lenvatinib or Bevacizumab in the Treatment of Subjects With Advanced Primary Liver Cancer
Brief Title: IBR900 Cell Injection Combined With Lenvatinib or Bevacizumab in the Treatment of Advanced Primary Liver Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Public Health Clinical Center (Other Government)
Collaborators: Imbioray (Hangzhou) Biomedicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBR900-T02
Record Dates: First submitted 2022-06-01; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Advanced Primary Liver Cancer
MeSH Terms: interventions — lenvatinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBR900 cell injection (Experimental): IBR900 Cell Injection Combined With Lenvatinib or Bevacizumab
  Interventions: Combination Product: IBR900 combined with Lenvatinib; Combination Product: IBR900 combined with Bevacizumab

INTERVENTIONS:
Combination Product: IBR900 combined with Lenvatinib — IBR900 cell injection: 4.0×10^9 cells, D1,D3 of each cycle. Lenvatinib: body weight ≥ 60kg, 12mg/qd; body weight < 60kg, 8mg/qd; administered continuously from D5 of the first cycle
Combination Product: IBR900 combined with Bevacizumab — IBR900 cell injection: 4.0×10^9 cells, D1,D3 of each cycle. Bevacizumab:15mg/kg, D1 of each cycle.

SUMMARY:
This is an open-label, nonrandomized investigator-initiated clinical trial to evaluate the safety, tolerability, and efficacy of IBR900 cell injection in combination with Lenvatinib or bevacizumab in subjects with advanced primary liver cancer.

DETAILED DESCRIPTION:
Two treatment groups are set up in this study. The first treatment group is IBR900 cell injection combined with Lenvatinib. The second treatment group is IBR900 cell injection combined with bevacizumab. Each cycle of the two treatment groups is 21 days. After 4 cycles of treatment, if the investigator judges that the subjects may benefit from continuing treatment, the subjects can continue to receive more cycles of treatment. 6 subjects are enrolled in each treatment group, and the group assignment of subjects is determined by the investigator.

For subjects who have previously received Lenvatinib, they will not be able to continue to receive Lenvatinib after entering the study, but can be treated in combination with bevacizumab. For subjects who have previously received bevacizumab, they will not be able to continue to receive bevacizumab after entering the study, but can be treated in combination with Lenvatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age≥18 and ≤75 years old.
2. Subjects with stage IIb, # or IV unresectable / advanced primary hepatocellular carcinoma, intrahepatic cholangiocarcinoma or mixed hepatocellular cholangiocarcinoma diagnosed in accordance with the Guidelines for Diagnosis and Treatment of Primary Liver Cancer of CSCO(2020 Edition).
3. Having ≥ 1 measurable lesion in accordance with the modified Response Evaluation Criteria in Solid Tumors (mRECIST) (lesions located in the field of previous radiation therapy cannot be used as target lesions unless there is imaging evidence that the lesion has progressed or persisted three months after radiation therapy).
4. Have a performance status of 0 or 2 on the ECOG Performance Score, life expectancy ≥12 weeks.
5. Male and female subjects of childbearing age and their partners must agree to take effective birth controls (hormone, barrier method or abstinence, etc.) from signing the ICF to 6 months after the last administration.
6. Subjects should voluntarily participate in this clinical study, are fully aware of the study, have signed the Informed Consent Forms, and are willing to follow and able to complete all trial procedures.

Exclusion Criteria:

1. Received systemic anti-tumor therapy within 4 weeks prior to the first administration, including chemotherapy, immunotherapy, radical radiotherapy, etc.; received palliative radiotherapy within 2 weeks prior to the first administration; or the adverse events caused by previous anti-tumor therapy have not recovered to ≤Grade 1 (except for alopecia).
2. Have known central nervous system metastases with clinical symptoms.
3. Received any adoptive cellular immunotherapy within 6 months prior to the first administration.
4. Have undergone major organ surgery (excluding needle biopsy or surgery related to this indication) within 4 weeks prior to their first administration of the study drug, or required elective surgery during the study period.
5. Have received or expected to receive glucocorticoids (prednisone >10 mg daily or equivalents) or other immunosuppressive medications within 14 days prior to the first administration. Note: For subjects without active autoimmune disorder, inhaled or topical steroid hormone or equivalent dose of prednisone ≤ 10 mg/day is allowed, and glucocorticoid is allowed for short-term (≤ 7 days) preventive treatment (e.g. contrast media allergy) or for the treatment of non-autoimmune disorder (e.g. delayed type hypersensitivity to contact allergens).
6. Received live or attenuated vaccine within 4 weeks prior to the first administration or plan to receive live or attenuated vaccine during the study period.
7. Patients with severe infections that cannot be controlled.
8. Patients with a known history of human immunodeficiency virus (HIV) active infection.
9. Have active autoimmune diseases or have had autoimmune diseases that are likely to recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, vasculitis, psoriasis, etc.). Except in the following cases: type 1 diabetes well controlled with hormone replacement therapy, hypothyroidism, skin conditions not requiring systemic therapy (such as vitiligo), and other conditions that are well controlled and that are less likely to relapse as by the investigator (such as resolved childhood asthma).
10. Organ function during screening should meet the following criteria:

    1. Absolute neutrophil count (ANC)<1.5×10^9/L, platelet (PLT)<75×10^9/L, hemoglobin (Hb)<80g/L, (blood transfusion, platelet and colony stimulating factor therapy are not allowed within 2 weeks before the test);
    2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)>5 times the upper limit of normal (ULN), and total serum bilirubin>2.5 times the upper limit of normal (ULN);
    3. Creatinine(Cr)>1.5×ULN, and creatinine clearance rate(Ccr) ≤ 60ml/min (estimated according to Cockcroft-Gault formula). Note: Ccr to be calculated only when Cr >1.5×ULN;
    4. International normalized ratio (INR) ≤ 2.0×ULN, activated partial thrombin time (APTT) >1.5×ULN.
11. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    1. There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia, and Ⅱ-Ⅲ degree atrioventricular block, which need clinical intervention;
    2. The mean QT interval corrected by Fridericia method (QTcF) is prolonged (male>450ms, female>470ms);
    3. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or above cardiovascular and cerebrovascular events occurring within 6 months before the first administration;
    4. Patients with heart failure or left ventricular ejection fraction (LVEF) < 50% in the New York Heart Association (NYHA) classification ≥II;
    5. Hypertension beyond clinical control;
12. Subjects with previous or current interstitial lung disease, pneumoconiosis, radiation pneumonia, severe impairment of pulmonary function that may interfere with the detection and treatment of suspected drug-related pulmonary toxicity. Or uncontrolled systemic diseases, including diabetes, etc.
13. Had other malignant tumors in the past 3 years, except for any type of carcinoma in situ that has been cured in the past and cured skin basal cell carcinoma or skin squamous cell carcinoma.
14. Pregnant women or lactating women.
15. Have a history of drug abuse.
16. Patients with a history of serious dementia, mental status changes or any history of mental disorder, incapacity or limited capacity.
17. Have participated in other clinical trials and received any unmarketed investigational drug or treatment within 4 weeks prior to the first administration.
18. Patients who have received anti-tumor treatment with lenvatinib and bevacizumab.
19. According to the judgment of the investigators, other factors that may make the subjects unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From day 1 to day 90 after the last infusion
  The incidence and severity of adverse events assessed according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0, and the correlation between adverse events and IBR900 cell injection.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year after infusion
  The proportion of subjects with complete and partial tumor remissions after treatment
Progression-free survival (PFS) | Up to 1 year after infusion
  The time from the beginning of treatment to the onset of tumor progression or death from any cause
Overall survival (OS) | Up to 5 year after infusion
  From the beginning of treatment to the time of death from any cause
Disease control rate (DCR) | Up to 1 year after infusion
  Proportion of subjects with complete, partial response and stable disease
Best of response (BOR) | Up to 1 year after infusion
  The rate of best of disease response recorded from the beginning of study treatment to disease progression, recurrence, or death.

OTHER OUTCOMES:
Cytokine release | Up to 1 year after infusion
  Blood samples will be collected at specified time points to detect the cytokine (IL-1β, IL-2, IL-4, IL-6, IL-10, IFN-γ, TNF-α) concentration
Lymphocyte subtype | Up to 1 year after infusion
  Blood samples will be collected at specified time points to analyze the lymphocyte subtypes (CD3, CD4, CD8, CD19, CD56)

CONTACTS AND LOCATIONS:
Overall Officials: Jingbo Wang, Principal Investigator — Head of the department of Biology and Cell therapy